CLINICAL TRIAL: NCT05326698
Title: Evoked Potential Response to Full-endoscopic Cervical Foraminotomy
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional de la Citadelle (Other)
Responsible Party: Principal Investigator, Remacle Thibault, MD, PhD, Neurosurgeon, Principal Investigator, Centre Hospitalier Régional de la Citadelle
Other Study IDs: Evoked cervical endoscopy
Record Dates: First submitted 2022-02-16; First posted 2022-04-13 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Cervical Foraminal Stenosis
Keywords: Evoked Potential; Endoscopy; Irrigation pressure; Dorsal columns

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Medtronic NIM Eclipse for evoked potentials recording — Recording of somesthetic and motor evoked potentials during endoscopic posterior cervical foraminotomy.
  Other Names: Joimax Ilessys Pro for endoscopic cervical foraminotomy

SUMMARY:
Cervical foraminotomy is used to treat recalcitrant foraminal stenosis in the cervical region. This foraminotomy can be performed under endoscopy. The irrigation pressure used to allow adequate visualization of the anatomical structures is usually between 40 and 50 mmHg. This pressure has no adverse effect intraoperatively on motor evoked potentials but its effect on somesthetic evoked potentials has not yet been studied. The purpose of this study is to validate the absence of disruption of somatosensory evoked potentials by endoscopic cervical foraminotomy

ELIGIBILITY:
Inclusion Criteria:

1. Cervical radiculopathy due to foraminal stenosis
2. Age > 18 years
3. Radicular arm pain that were refractory to optimal medical therapy for a minimum of 3 months.
4. Persistent pain despite 3 types of pharmacological treatments (paracetamol, non-steroidal anti-inflammatory drugs, opioids, antidepressant medications, and anticonvulsant medications, etc.).
5. Intact Llemniscal pathways must remain at least partially intact

Exclusion Criteria:

1. History of coagulation disorders; Lupus erythematosus; diabetic neuropathy; rheumatoid arthritis; Morbus Bechterew; Active malignancy; immune deficiency
2. Presence of myelopathy
3. Addiction to drugs, alcohol (5 units/day) and/or medications

Age Groups: Child, Adult, Older Adult
Study Population: 3 patients will undergo endoscopic surgery on February 22 and 23, 2022 for a cervical foraminotomy to treat foraminal stenosis responsible for recalcitrant cervicobrachial pain. These surgeries will be performed with pre-, per- and post-operative recording of motor and sensory evoked potentials.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2022-02-22 (Actual); Primary Completion 2022-02-23 (Actual); Study Completion 2022-02-24 (Actual)

PRIMARY OUTCOMES:
Influence of the endoscopic irrigation pressure on somatosensory evoked potentials. | Through surgery completion, from electrodes placement until their removal. An average of two hours.
  The evoked potentials electrodes were placed once the patient was asleep under general anesthesia, installed in a prone position in a Mayfield head holder.
  The electrodes were removed at the end of surgery after skin closure but before removing the headrest and returning the patient to his back.
  Somatosensory evoked potentials (SEP) were recorded continuously from electrode placement to electrode removal.
  The blood pressure and the irrigation pressure in the endoscope are also continuously recorded.
  A change SEP in latency and/or amplitude could therefore be detected during the entire recording and related to variations in irrigation pressure and intraoperative events.
Influence of the endoscopic irrigation pressure on motor evoked potentials. | Through surgery completion, from electrodes placement until their removal. An average of two hours.
  The evoked potentials electrodes were placed once the patient was asleep under general anesthesia, installed in a prone position in a Mayfield head holder.
  The electrodes were removed at the end of surgery after skin closure but before removing the headrest and returning the patient to his back.
  Motor evoked potentials (MEP) were recorded at each step of the surgery (preoperative, skin incision, working tube placement, endoscope introduction, and foraminotomy) and also at each variation of the irrigation pressure.
  A change MEP amplitude could therefore be detected during the entire recording and related to variations in irrigation pressure and intraoperative events.

CONTACTS AND LOCATIONS:
Locations (1):
- CHR Citadelle, Liège, Belgium

IPD SHARING:
Plan to Share IPD: Undecided